CLINICAL TRIAL: NCT03870230
Title: Investigation of Neurovascular Coupling in Glaucoma Patients and Healthy Subjects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Principal Investigator, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OPHT-010213
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-04

CONDITIONS: Glaucoma, Open-Angle; Normal Tension Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Low Tension Glaucoma; Ocular Hypertension | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- POAG MD<10dB (Experimental): patients with primary open angle glaucoma with MD in visual field less than or equal 10dB
  Interventions: Device: Fourier Domain Doppler Optical Coherence Tomography (FDOCT); Device: Dynamic Vessel Analyzer (DVA); Device: Pattern Electroretinography (pERG); Device: Optical coherence tomography (OCT); Device: Laser Speckle Flowgraphy (LSFG)
- POAG MD>10dB (Experimental): patients with primary open angle glaucoma with MD in visual field more than 10dB
  Interventions: Device: Fourier Domain Doppler Optical Coherence Tomography (FDOCT); Device: Dynamic Vessel Analyzer (DVA); Device: Pattern Electroretinography (pERG); Device: Optical coherence tomography (OCT); Device: Laser Speckle Flowgraphy (LSFG)
- NTG MD<10dB (Experimental): patients with normal tension glaucoma with MD in visual field less than or equal 10dB
  Interventions: Device: Fourier Domain Doppler Optical Coherence Tomography (FDOCT); Device: Dynamic Vessel Analyzer (DVA); Device: Pattern Electroretinography (pERG); Device: Optical coherence tomography (OCT); Device: Laser Speckle Flowgraphy (LSFG)
- NTG MD>10dB (Experimental): patients with normal tension glaucoma with MD in visual field more than 10dB
  Interventions: Device: Fourier Domain Doppler Optical Coherence Tomography (FDOCT); Device: Dynamic Vessel Analyzer (DVA); Device: Pattern Electroretinography (pERG); Device: Optical coherence tomography (OCT); Device: Laser Speckle Flowgraphy (LSFG)
- OHT (Experimental): patients with ocular hypertension
  Interventions: Device: Fourier Domain Doppler Optical Coherence Tomography (FDOCT); Device: Dynamic Vessel Analyzer (DVA); Device: Pattern Electroretinography (pERG); Device: Optical coherence tomography (OCT); Device: Laser Speckle Flowgraphy (LSFG)
- controls (Experimental): healthy, age and sex matched, control subjects
  Interventions: Device: Fourier Domain Doppler Optical Coherence Tomography (FDOCT); Device: Dynamic Vessel Analyzer (DVA); Device: Pattern Electroretinography (pERG); Device: Optical coherence tomography (OCT); Device: Laser Speckle Flowgraphy (LSFG)

INTERVENTIONS:
Device: Fourier Domain Doppler Optical Coherence Tomography (FDOCT) — Retinal blood flow will be assessed using FDOCT
Device: Dynamic Vessel Analyzer (DVA) — Retinal vessel diameters and oxygen saturation will be measured with the DVA device
Device: Pattern Electroretinography (pERG) — to assess the neuronal function of the retina, pattern ERG will be performed
Device: Optical coherence tomography (OCT) — to assess the morphology of the retina, OCT will be performed
Device: Laser Speckle Flowgraphy (LSFG) — to assess retinal blood flow, LSFG will be performed

SUMMARY:
Glaucoma is characterized by a progressive loss of retinal ganglion cells (RGCs) leading to optic nerve head (ONH) damage and associated visual field defects. The main risk factor for glaucoma is elevated intraocular pressure (IOP). Reducing IOP slows down the progression of the disease as several large multicenter trials have shown. Some patients, however, still progress despite adequately controlled IOP. As such, there is considerable interest in approaches that rescue RGCs independent of IOP, a strategy called neuroprotection. Although this field was actively discovered in the last 20 years in the brain and the eye, no non-IOP related treatment is clinically available to date. Various approaches are currently studied in some detail. One interesting strategy focuses on the neurovascular unit.

The blood flow of the human retina is controlled by complex mechanisms that include myogenic, metabolic and hormonal factors. The high consumption of oxygen in the human retina is crucial for normal functioning of the organ. As in the brain, blood flow in the retina is also controlled by neurovascular coupling. This means that the retina increases its blood flow to regions in which neurons are activated. This is done in an effort to provide more oxygen and glucose to the active neurons. In the recent years evidence has accumulated that astrocytes play a key role in mediating this vasodilator signal.

In the brain, abnormalities in neurovascular coupling have been observed in diseases like stroke, hypertension, spinal-cord injury and Alzheimer's disease. This break-down of neurovascular coupling is considered to play a key role in neuronal death in these diseases. In the retina, abnormalities in neurovascular coupling have been observed in diseases as diabetes and glaucoma.

Most of the data obtained in the human retina stem from a system that measures retinal vasodilatation during stimulation with flickering light. The investigators have previously shown that flicker stimulation of the retina is, however, also associated with a pronounced increase in retinal blood velocities. In this study the investigators employed laser Doppler velocimetry (LDV) for the measurement of retinal blood velocities, but this technique is not clinically applicable because it requires excellent fixation of the subject under study. In the present study, the investigators propose to use an alternative system for neurovascular coupling that they have developed recently. In this approach, the investigators use bi-directional Fourier-domain optical coherence tomography for the assessment of retinal blood flow. Optical coherence tomography (OCT) is a non-invasive optical imaging modality enabling cross-sectional tomographic in vivo visualization of internal microstructure in biological systems. In ophthalmology, OCT has become a standard tool in visualizing the retina and nowadays is considered also as a standard tool in the diagnosis of retinal disease. In the recent years, conventional time domain OCT was replaced by Fourier domain OCT providing significantly improved signal quality.

This bidirectional system overcomes the limitations of previously realized techniques, which include doubtful validity and limited reproducibility. In addition, pattern ERG, multifocal ERG and oscillatory potentials will be measured to allow for concomitant assessment of neural function.

The investigators seek to measure neurovascular coupling in the human retina in patients with early primary open angle glaucoma (POAG), normal tension glaucoma, ocular hypertension and a healthy control group. In order to obtain information on neurovascular coupling, both neuronal function as well as retinal blood flow need to be measured. In the present study, the investigators will employ pattern ERG, multifocal ERG as well as oscillatory potentials to assess the function of the inner retina. Retinal blood flow through major retinal arterial and venous branch vessels will be measured before, during and after flicker stimulation with the dual-beam bidirectional Fourier Domain Doppler OCT coupled to the commercially available Dynamic Vessel Analyzer (DVA) produced by IMEDOS, Jena, Germany, which provides adequate resolution to study the retinal circulation.

ELIGIBILITY:
Inclusion criteria

Patients with primary open angle glaucoma

* Diagnosis of manifest primary open angle glaucoma defined as pathological optic disc appearance
* Glaucoma hemifield test outside normal limits
* Untreated IOP ≥ 21 mmHg on at least three measurements in the medical history
* Mean deviation in the visual field test is less than or equal 10dB (for one group) OR more than 10dB (for the other group)

Patients with normal tension glaucoma

* Diagnosis of manifest normal tension glaucoma defined as pathological optic disc appearance
* Glaucoma hemifield test outside normal limits
* No evidence of untreated IOP > 20 mmHg in the medical history
* Mean deviation in the visual field is less than or equal 10dB (for one group) OR more than 10dB (for the other group)

Patients with ocular hypertension

* Normal ophthalmic findings except presence of ocular hypertension defined as untreated IOP ≥ 21 mmHg on at least three measurements in the medical history
* No signs of glaucomatous damage in the optic disc
* or the glaucoma hemifield test

Healthy control subjects

* Normal ophthalmic findings
* IOP < 20 mmHg on least three measurements
* No evidence of increased IOP in the medical history
* No signs of glaucomatous damage in the optic disc
* or the glaucoma hemifield test

Exclusion criteria

* History of a severe medical condition as judged by the clinical investigator
* Abuse of alcoholic beverages
* Smoker
* Participation in a clinical trial in the 3 weeks preceding the study
* Exfoliation glaucoma, pigmentary glaucoma, history of acute angle closure
* Intraocular surgery within the last 6 months
* Ocular inflammation or infection within the last 3 months
* History of epilepsia
* Diabetes mellitus
* Untreated hypertension with systolic blood pressure > 160 mmHg, diastolic blood pressure > 95 mmHg
* Pregnancy
* Planned pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Flicker induced blood flow alterations | 1 day
  Response of retinal blood flow to flicker light

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhöfer, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No